CLINICAL TRIAL: NCT00461877
Title: High-Risk HPV Infections in Women Aged 25 to 65
Status: Completed | Type: Observational
Sponsor: University of Washington (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Rachel Winer, Assistant Professor, University of Washington
Other Study IDs: 31286
Record Dates: First submitted 2007-04-16; First posted 2007-04-18 (Estimated); Last update posted 2013-11-19 (Estimated); Status verified 2013-11

CONDITIONS: Papillomavirus Infections
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Vaginal swab samples for HPV DNA testing
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine risk factors for HPV infections in 25 to 65 year old women who report having used internet dating websites in the past year.

DETAILED DESCRIPTION:
Whether older women are susceptible to acquiring new, persistent high-risk (HR) HPV infections from new sex partners is largely unknown. This is a pilot study of predictors of HR HPV infections in two populations of women aged 25 to 44 and 45 to 65 who have used internet dating websites in the past year. 400 women will be recruited and mailed kits for self-collecting vaginal specimens for HPV DNA testing. Women will self-collect two sets of vaginal specimens four months apart, and complete sexual behavior questionnaires at the time of each self-collection. If new HPV infections associated with recent new partners are detected in these women, this pilot data will be used to develop a larger longitudinal study of the acquisition and natural history of HR HPV infections in older women. This information is important for developing guidelines for HPV vaccine implementation and cervical cancer screening guidelines in populations of older women.

ELIGIBILITY:
Inclusion Criteria:

* Have had sex with men
* Have used the internet to search for romantic partners in the past year (e.g. posted or responded to an ad on an internet dating website or social networking website)

Exclusion Criteria:

* Pregnant, breastfeeding, or planning a pregnancy in the next 6 months
* Hysterectomy

Ages: 25 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 25 to 65 year old women who date online
Sampling Method: Non-Probability Sample
Enrollment: 303 (Actual)
Dates: Start 2007-03; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
High-Risk HPV DNA | four months

CONTACTS AND LOCATIONS:
Overall Officials: Rachel L Winer, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

REFERENCES:
- See also: HPV study website — http://depts.washington.edu/hpvstudy